CLINICAL TRIAL: NCT07283536
Title: Two-site Blind Epidural Patch Versus Targeted Epidural Patch With Autologous Platelet-rich Plasma for Spontaneous Intracranial Hypotension: A Prospective, Assessor Blind, Randomized, Controlled, Noninferiority Trial
Brief Title: Blind Versus Targeted Epidural Patch With Autologous Platelet-rich Plasma for Spontaneous Intracranial Hypotension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2023-263-03-08
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Spontaneous Intracranial Hypotension
MeSH Terms: conditions — Intracranial Hypotension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blind epidural PRP patch (BEPP) (Experimental): Two-site blind epidural patch with PRP, which was prepared with the 2-stage centrifugation method, at levels C7-T1 and L4-5.
  Interventions: Procedure: Blind epidural PRP patch
- Targeted epidural PRP patch (TEPP) (Active Comparator): Targeted epidural patch with autologous platelet-rich plasma, which was prepared with the 2-stage centrifugation method.
  Interventions: Procedure: Targeted epidural PRP patch

INTERVENTIONS:
Procedure: Targeted epidural PRP patch — Each patient was subjected to either magnetic resonance myelography (MRM) or/and computed tomography myelography (CTM) to detect the location of CSF leaking. PRP was prepared with the 2-stage centrifugation method and a standard epidural puncture was conducted at the definitive CSF leak locations under the guidance of CT. A predetermined volume of PRP (no more than 10 mL) was titrated slowly into the epidural space for each level. A strict bed stay for 48 h was prescribed in supine position postoperatively.
  Arms: Targeted epidural PRP patch (TEPP)
Procedure: Blind epidural PRP patch — PRP was prepared with the 2-stage centrifugation method and the investigators chose two separate sites for epidural access, the C7-T1 and L4-5 levels. A standard epidural puncture was conducted under the guidance of CT. A predetermined volume of PRP (no more than 10 mL) was titrated slowly into the epidural space for each level. A strict bed stay for 48 h was prescribed in supine position postoperatively.
  Arms: Blind epidural PRP patch (BEPP)

SUMMARY:
Spontaneous intracranial hypotension (SIH) is a condition characterized by refractory orthostatic headache, mostly due to loss of cerebrospinal fluid (CSF). Epidural patch with autologous platelet-rich plasma (PRP), which contains numerous growth factors and cytokines, has been reported as a successful alternative for whole blood in dura repair. However, there is no report regarding the best approach to use: targeted epidural PRP patch (TEPP) versus blind epidural PRP patch (BEPP). Preliminary work has suggested that both targeted and blind approaches are effective when using whole blood for epidural patch. Furthermore, two-site blind approach could be considered as a viable initial treatment regardless of the identification of the leak for conventional targeted approach. In this study, the investigators aimed to investigate the non-inferiority of two-site BEPP compared with TEPP for the treatment of refractory SIH cases failing in conservative therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent to participate the research obtained from the patient.
2. Age 18-65 years.
3. Satisfies the criteria for SIH according to the International Classification of Headache Disorders criteria for headaches attributed to spontaneous (or idiopathic) low CSF pressure.
4. Failed conservative management (bed rest oral or intravenous hydration, and analgesics) lasting at least 2 weeks.

Exclusion Criteria:

1. There was concern for other causes of intracranial hypotension, such as postdural puncture, postsurgical and post-traumatic CSF leaks.
2. Prior treatment with EBP at any time previously.
3. Any contraindication to epidural puncture, such as space-occupying intracranial or intraspinal lesions, spinal defect, suspected infection over the puncture site, bleeding disorder and current anticoagulation therapy.

   History of drug and alcohol abuse, cognitive dysfunction, or mental illness.
4. Unable to comprehend the pain NRS.
5. Unable to cooperate with postoperative treatment, rehabilitation, and follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain NRS of orthostatic headache | 48 hours following epidural patch with PRP
  Pain intensity was evaluated by pain numeric rating scale (NRS; 0 = no pain, 10 = unbearable pain) for headache.

SECONDARY OUTCOMES:
Pain NRS of orthostatic headache | 1, 3 and 6 months following epidural patch with PRP
  Pain intensity was evaluated by pain numeric rating scale (NRS; 0 = no pain, 10 = unbearable pain) for orthostatic headache .
The complete relief rate of epidural patch with PRP | 48 hours, 1, 3 and 6 months after the initial targeted or blind patch
  The complete relief was defined as the pain intensity of 0-1/10 on NRS or/and minimal symptoms post-procedurally.
The good response rate of epidural patch with PRP | 48 hours, 1, 3 and 6 months post-procedurally
  Good response was defined as a headache reduction of at least 50%, with improvement of orthostatic component post-procedurally.
The failure rate of epidural patch with PRP | 48 hours following the initial epidural patch with PRP
  Failure was defined as a persistent or worsening symptom with less than 50% of headache reduction within 48 hours following the initial epidural patch with PRP
The recurrence rate in each group. | During the 6-month follow up
  Recurrence was defined as fresh onset of headaches beyond the 72-hour mark.
Patients' overall satisfaction | 6 months following the first epidural patch with PRP
  Patients' overall satisfaction was graded into very unsatisfactory (1), unsatisfactory (2), neutral (3), satisfactory (4) and very satisfactory (5), according to the Likert scale.
The occurrence of complications | During and after the epidural patch with PRP until the end of 6-month follow up
The percent of patients requiring repeat epidural PRP patch | During the 6- month follow up

IPD SHARING:
Plan to Share IPD: Undecided